CLINICAL TRIAL: NCT06857422
Title: Effect of Hand Fan Applied to COPD Patients on Dyspnea, Illness Perception, Anxiety and Depression: A Double-Blind Randomized Controlled Experimental Study
Brief Title: Dyspnea and Psychosocial Effects of Hand Fan Application in COPD Patients
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ardahan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ArdahanU-Simsekli-DS-04
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: COPD; Dyspnea; Illness Perception; Anxiety; Depression
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Anxiety Disorders; Depression | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding will be done for the researcher, participants and statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): hand fan application
  Interventions: Behavioral: Hand Fan Application
- Control group (Active Comparator): standard care
  Interventions: Other: Standard Care for COPD Patients

INTERVENTIONS:
Behavioral: Hand Fan Application — Participants in the experimental group will be instructed to use a hand fan to cool their face for 10 minutes each day for a period of 6 weeks. The fan should be held approximately 15 cm from the face, focusing on the middle area. This intervention aims to alleviate symptoms of dyspnea and improve psychological well-being, including anxiety, depression, and illness perception. The participants will receive daily reminders to ensure consistent application of the intervention.
  Arms: Experimental group
Other: Standard Care for COPD Patients — Participants in the control group will receive standard care for chronic obstructive pulmonary disease (COPD) patients. This includes routine management and treatment as prescribed by their healthcare providers, such as medication and lifestyle recommendations. They will not be instructed to use a hand fan or any other cooling device during the study period. The control group will continue their regular care without any additional interventions from the research team.
  Arms: Control group

SUMMARY:
This randomized controlled trial aims to evaluate the effects of hand fan application on dyspnea, illness perception, anxiety, and depression in COPD patients. A total of 56 voluntary COPD patients (28 experimental, 28 control) will be recruited from Ardahan State Hospital Chest Diseases Clinic.

Patients will be randomly assigned to the experimental or control group. The experimental group will receive a hand fan and use it for 10 minutes daily for six weeks, while the control group will receive standard care. Dyspnea, illness perception, anxiety, and depression will be assessed using the Visual Dyspnea Scale, Illness Perception Questionnaire, and Hospital Anxiety and Depression Scale at baseline and after six weeks.

Data will be analyzed using statistical software. This study is expected to contribute to the literature by evaluating a non-pharmacological intervention for COPD-related dyspnea and psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Orientation and cooperation
* No communication problems

Exclusion Criteria:

* Having a COPD exacerbation in the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-14 (Actual)

PRIMARY OUTCOMES:
Dyspnea Severity | Pre-intervention: Before the start of the intervention (baseline measurement).Post-intervention: After 6 weeks of intervention (final measurement).
  The primary outcome measure of this study will be the severity of dyspnea, assessed using the Visual Analog Scale (VAS). This scale is a subjective tool used to measure the intensity of shortness of breath experienced by participants.

SECONDARY OUTCOMES:
Illness Perception | Pre-intervention: Before the start of the intervention (baseline measurement).Post-intervention: After 6 weeks of intervention (final measurement).
  Measured using the Illness Perception Questionnaire
Anxiety and Depression | Pre-intervention: Before the start of the intervention (baseline measurement).Post-intervention: After 6 weeks of intervention (final measurement).
  Measured using the Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Locations (1):
- Derya ŞİMŞEKLİ, Ardahan, Ardahan, Turkey (Türkiye)